CLINICAL TRIAL: NCT03602950
Title: Role of Autologous Platelet-Rich Plasma Solution in Wound Healing in Diabetic Patients Undergoing Elective Cesarean Delivery
Brief Title: PRP Use in Diabetic Patients Undergoing Cesarean Section
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hany Hassan Kamel, principal investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MiniaU2018
Record Dates: First submitted 2018-07-06; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Diabetes, Gestational; Wound Complication
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: The intervention group will receive PRP at surgery, whereas the control group will receive the usual care. All patients will be evaluated at baseline, one week, four weeks and eight week after the cesarean section.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): 50 diabetic ladies at full term will undergo elective CS and will receive the usual surgical care routinely done at our hospital
- study group (Active Comparator): 50 diabetic ladies will undergo elective CS at full term and autologous PRP will be injected subcutaneously before skin closure.
  Interventions: Biological: PRP

INTERVENTIONS:
Biological: PRP — autologous PRP will be injected subcutaneously before skin closure at time of elective CS
  Arms: study group

SUMMARY:
this study will investigate the effectiveness of PRP in wound healing among diabetic patients undergoing elective cesarean sections

DETAILED DESCRIPTION:
In this balanced, randomized, and controlled prospective study, 100 pregnant ladies at full term diabetic patients will be admitted to Minia University hospital. The patients will be randomly assigned into two groups. The intervention group will receive PRP at surgery, whereas the control group will receive the usual care. All patients will be evaluated at baseline, one week, two weeks, four weeks and eight week after the cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be a fixed factor along with age(18 y:45 y),diabetic patients(any type of diabetes),elective delivery,average body mass index(BMI) (17 : 24.9),Non previously scared uterus ,single pregnancy

Exclusion Criteria:

* The exclusion criteria will be younger ages below 18 years ,older ages above 45 years, emergency caesarean delivery, previous scared uterus, underweight BMI below 17, overweight BMI above 24.9, no other medical problems, associated other diseases, and multiple pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
changes in wound healing | one week post-operatively
  REEDA descriptive scale will assess degree of wound healing which formed of 4 points in a categorical score assessing 5 items of healing, redness, edema,ecchymosis,discharge ,approximation of the wound edges. each item is rated on a scale of 0-3 and total score may range between 0-15. lower scores indicating good healing

SECONDARY OUTCOMES:
morbidly wound healing | 4-8weeks
  at 4 and 8 weeks post-operatively the wound healing will be completed and will be assessed using VSS,Vancouver scar scale, which detect formation of keloid or hypertrophic scars. it will assess vascularity, scar thickness, pliability and pigmentation

IPD SHARING:
Plan to Share IPD: No